CLINICAL TRIAL: NCT04006678
Title: Evaluation of Accuracy of Computer Guided Versus Conventional Segmental Sandwich Osteotomy With Immediate Implant Placement in Vertically Deficient Anterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shareif Qassim Shareif Nazzal, ORAL & MAXILLOFACIAL SURGERY MASTER CANDIDATE, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-18-06-2019
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Sandwich Osteotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided sandwich osteotomy (Experimental): segmental sandwich osteotomy will be done for vertically deficient ridges in anterior area of the maxilla. Either using surgical guides (Computer guide segmental sandwich osteotomy technique) for study group and conventional segmental sandwich osteotomy technique for control group.
  Interventions: Procedure: computer guided sandwich osteotomy
- conventional sandwich osteotomy (Active Comparator): :conventional segmental sandwich osteotomy will be done for vertically deficient ridges in anterior area of the maxilla.
  Interventions: Procedure: computer guided sandwich osteotomy

INTERVENTIONS:
Procedure: computer guided sandwich osteotomy — segmental sandwich osteotomy will be done for vertically deficient ridges in anterior area of the maxilla. Either using surgical guides (Computer guide segmental sandwich osteotomy technique) for study group and conventional segmental sandwich osteotomy technique for control group.

SUMMARY:
In conventional segmental sandwich osteotomy technique the moving the transport segment inferiorly to increase the vertical height causes the segment to move bucco-palatally, increasing the horizontal defect. So using the computer guided in segmental sandwich osteotomy and fixation the transport segment hopefully will reduce the bucco-palatal tipping.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vertically deficient anterior maxillary ridge a minimum 10 mm. height of alveolar bone.
* Patients with medical history that did not hinder implant placement (uncontrolled diabetes) and adequate proper oral hygiene.
* Patients of adequate alveolar bone width.
* Both genders males and females will be included.

Exclusion Criteria:

* General contraindications to implant surgery.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Lack of opposite occluding dentition/prosthesis in the area intended for implant placement.
* Active infection or severe inflammation in the area intended for implant placement.
* Need of bone augmentation procedures at implant placement.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly followed.
* Referred only for implant placement or unable to attend a 5-year follow-up.
* Requiring only single implant-supported crowns.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
bucco - palatal tipping | 6 months
  calculate the amount of bucco-palaltal tipping of mobilized transport segment after 6 months in mm by cone beam CT between both groups.

SECONDARY OUTCOMES:
marginal bone loss | 6 months
  calculate marginal bone loss in mm by cone beam CT between two groups

CONTACTS AND LOCATIONS:
Overall Officials: shareif nazzal, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided